CLINICAL TRIAL: NCT01896245
Title: Laryngeal Injuries After Anesthesia Induction With Three Different Sevoflurane Concentrations (Without Muscle Relaxant)
Acronym: SEVODosage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, Clinical Associate Professor Dr Thomas Mencke, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A 2013-0039
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Other Specified Injuries of Vocal Cord, Sequela
Keywords: hoarseness; sore throat; intubating conditions; vocal cord injuries; sevoflurane
MeSH Terms: conditions — Hoarseness; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sevoflurane 1,0 (Active Comparator): sevoflurane 1,0: sevoflurane is administered with a concentration of 1,0 MAC
  Interventions: Drug: sevoflurane 1,0
- sevoflurane 1,2 (Active Comparator): sevoflurane 1,2: sevoflurane is administered with a concentration of 1,2 MAC
  Interventions: Drug: sevoflurane 1,2
- sevoflurane 1,4 (Active Comparator): sevoflurane 1,4: sevoflurane is administered with a concentration of 1,4 MAC
  Interventions: Drug: sevoflurane 1,4

INTERVENTIONS:
Drug: sevoflurane 1,0 — anesthesia induction with propofol, remifentanil, and sevoflurane 1,0 MAC; afterwards tracheal intubation
  Other Names: sevo 2,0 %
  Arms: sevoflurane 1,0
Drug: sevoflurane 1,2 — anesthesia induction with propofol, remifentanil, and sevoflurane 1,2 MAC; afterwards tracheal intubation
  Other Names: sevo 2,5 %
  Arms: sevoflurane 1,2
Drug: sevoflurane 1,4 — anesthesia induction with propofol, remifentanil, and sevoflurane 1,4 MAC; afterwards tracheal intubation
  Other Names: sevo 3,0 %
  Arms: sevoflurane 1,4

SUMMARY:
Anesthesia induction and tracheal intubation can be performed with and without neuromuscular blocking agents (NMBAs). Tracheal intubation can be performed with sevoflurane instead of NMBAs; intubating conditions are similar and the incidence of vocal cord injuries are similar, too.

DETAILED DESCRIPTION:
We perform tracheal intubation with propofol, remifentanil and sevoflurane; sevoflurane is administered with three dosages. During tracheal intubation intubating conditions are noted. After surgery, all patients are examined by video laryngoscopy; moreover all patients are asked for hoarseness and sore throat.

ELIGIBILITY:
Inclusion Criteria:

* ear-nose-throat surgery
* orotracheal intubation for surgery of the ear
* ASA I-III

Exclusion Criteria:

* obesity
* allergy against the study drugs
* patients with a known or suspected difficult airway
* diseases of the larynx

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
incidence of vocal cord injuries | 24 hours after tracheal intubation

SECONDARY OUTCOMES:
incidence of hoarseness | 24, 48, and 72 hours after tracheal intubation
incidence of soar throat | 24, 48, and 72 hours after tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mencke, Dr., Principal Investigator — Dep. of Anesthesia and Intensive Care Medicine, University of Rostock, Germany
Locations (1):
- Department of Anesthesia and Intensive Care Medicine, University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Ovari A, Bicker I, Machmueller S, Schuldt T, Sauer M, Soltesz S, Noeldge-Schomburg G, Mlynski R, Mencke T. Sevoflurane at 1.0 MAC together with remifentanil and propofol produces clinically acceptable intubation conditions at the vocal cords: A prospective randomized study. J Int Med Res. 2017 Jun;45(3):1098-1108. doi: 10.1177/0300060517701355. Epub 2017 Apr 28. PMID 28449630